CLINICAL TRIAL: NCT00766571
Title: Clinical and Genetic Studies of VACTERL Association
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080224; 08-HG-0224
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2017-06-29

CONDITIONS: Congenital Abnormalities; Birth Defects; Congenital Defects
Keywords: VACTERL Association; VATER Association; Multiple Congenital Anomalies; VACTERL; Congenital Defects; Birth Defects; Congenital Abnormalities
MeSH Terms: conditions — Congenital Abnormalities; VACTERL association; VATER association; Abnormalities, Multiple

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study will explore the medical problems in patients with VACTERL association and identify gene changes that might be responsible for them. VACTERL association can affect many parts of the body, including the bones of the spine, the heart, the lower intestinal tract, the connection between the trachea and esophagus, the kidneys and the arms. Information from this study may lead to a better understanding of the disease and improved treatment and genetic counseling.

Patients with VACTERL association and their parents and siblings may be eligible for this study.

Patients are admitted to the NIH Clinical Center for evaluation over 3 to 4 days that may include the following procedures:

* Physical examination, medical history, electrocardiogram (EKG), blood and urine tests
* Eye examination
* Imaging studies (echocardiogram, x-rays and ultrasound tests)
* Other specialized tests or consultations as indicated
* Optional medical photographs of the face and other body parts that may be involved in VACTERL association for publication in scientific texts or for teaching purposes
* Optional return visit after 2 years for repeat testing and to look for changes over time

Parents of patients have the following procedures:

* Physical examination, medical history, blood tests and x-rays, if needed
* Specialty consultations as indicated
* Optional medical photographs of the face and other body parts that may be involved in VACTERL association for publication in scientific texts or for teaching purposes
* Questionnaires about their child s medical history, growth, behavior and development, therapy and medication

Siblings of patients have the following procedures:

* Physical examination, medical history and blood tests

DETAILED DESCRIPTION:
The combination of vertebral defects, anal atresia, cardiac anomalies, tracheo-esophageal fistula, radial dysplasia and limb anomalies, and renal anomalies, termed VACTERL association, has been used as a clinical descriptor for a specific group of phenotypic manifestations that have been observed to occur together. Depending upon the diagnostic criteria used, the prevalence may be as high as 1 in 6000 live births. VACTERL association is felt to be due to defects in early embryogenesis, and is likely to be genetically heterogeneous. The purpose of the present study is to increase the understanding of the clinical manifestations and genetic causes of VACTERL association through detailed physical, laboratory, and radiological studies. We also plan to examine the spectrum of clinical characteristics in VACTERL association to facilitate early diagnosis and clinical management, including genetic counseling. To accomplish this, we plan to enroll approximately 25-50affected individuals along with their family members for a total of 75-150 total individuals each year, with an enrollment ceiling of 500 affected individuals. Patients and their families will be seen at the NIH clinical center.

ELIGIBILITY:
* INCLUSION CRITERIA:

(A) For affected individuals, determination of clinical criteria for inclusion will be determined by prior medical record review before participation. Inclusion criteria may be met in 1 of 3 ways:

1. At least 3 features of VACTERL association in an index case OR
2. Two features of VACTERL association in an index case plus at least 1 feature of VACTERL association in a relative OR
3. At least 2 features of VACTERL association in an index case plus at least 1 other anomaly.

(B) First degree relatives (parents and/or siblings of affected individuals) of patients with VACTERL association are also eligible to participate in portions of the protocol even if they have no features of VACTERL association.

EXCLUSION CRITERIA:

1. Anyone unwilling to provide informed consent (for themselves as adults, or on behalf of their children as minors, or on behalf of an adult who is unable to provide consent for themselves) or assent.
2. Cases that are clearly not in the spectrum of VACTERL association or related to our direct research interests (e.g. referred VACTERL cases that are felt to be related to other syndromes, such as Feingold syndrome, Townes-Brocks syndrome, or Pallister-Hall syndrome, would not be included). In such instances, we would attempt to make referrals to a more appropriate investigator.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2008-09-29; Study Completion 2017-06-29

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Muenke, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Arsic D, Beasley SW, Sullivan MJ. Switched-on Sonic hedgehog: a gene whose activity extends beyond fetal development--to oncogenesis. J Paediatr Child Health. 2007 Jun;43(6):421-3. doi: 10.1111/j.1440-1754.2007.01104.x. PMID 17535169
- [Background] Arsic D, Qi BQ, Beasley SW. Hedgehog in the human: a possible explanation for the VATER association. J Paediatr Child Health. 2002 Apr;38(2):117-21. doi: 10.1046/j.1440-1754.2002.00813.x. PMID 12030989
- [Background] Botto LD, Khoury MJ, Mastroiacovo P, Castilla EE, Moore CA, Skjaerven R, Mutchinick OM, Borman B, Cocchi G, Czeizel AE, Goujard J, Irgens LM, Lancaster PA, Martinez-Frias ML, Merlob P, Ruusinen A, Stoll C, Sumiyoshi Y. The spectrum of congenital anomalies of the VATER association: an international study. Am J Med Genet. 1997 Jul 11;71(1):8-15. doi: 10.1002/(sici)1096-8628(19970711)71:13.0.co;2-v. PMID 9215761